CLINICAL TRIAL: NCT00835666
Title: A Relative Bioavailability Study of Finasteride 5 mg Tablets Under Fasting Conditions
Brief Title: Finasteride 5 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: B026535
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Results first posted 2009-08-04 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Finasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Finasteride (Experimental): Finasteride 5 mg Tablet (test) dosed in first period followed by Proscar® 5 mg Tablet (reference) dosed in second period
  Interventions: Drug: Finasteride 5 mg tablets
- Proscar® (Active Comparator): Proscar® 5 mg Tablet (reference) dosed in first period followed by Finasteride 5 mg Tablet (test) dosed in second period
  Interventions: Drug: PROSCAR®

INTERVENTIONS:
Drug: Finasteride 5 mg tablets — 1 x 5 mg, single dose fasting
  Arms: Finasteride
Drug: PROSCAR® — 1 x 5 mg, single dose fasting
  Arms: Proscar®

SUMMARY:
The objective of this study is to compare the relative bioavailability of finasteride 5 mg tablets (manufactured and distributed by TEVA Pharmaceuticals USA) with that of PROSCAR® 5 mg tablets (Merck) in healthy, adult, non-smoking, male subjects under fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* All subjects selected for this study will be male non-smokers at least 18 years of age. Subjects will have a BMI (body mass index) of 30 or less.
* Each subject shall be given a general physical examination within 28 days of initiation of the study. Such examination includes, but is not limited to, blood pressure, general observations, and history.

Adequate blood and urine samples should be obtained within 28 days before beginning of the first period and at the end of the trial for clinical laboratory measurements.

Clinical laboratory measurements will include the following:

* Hematology: hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count (with differential).
* Clinical Chemistry: creatinine, BUN, glucose, SGOT/AST, SGPT/ALT, bilirubin, and alkaline phosphatase.
* Urine Analysis: pH, specific gravity, protein, glucose, ketones, bilirubin, occult blood, and cells.
* HIV Screen: pre-study
* Hepatitis B, C Screen: pre-study
* Drugs of Abuse Screen: pre-study and at each check-in Subjects will be selected if all above are normal. Electrocardiograms of all participating subjects will be recorded before initiation of the study and filed with each subject's case report forms.

Exclusion Criteria:

* Subjects with a history of chronic alcohol consumption (during past 2 years), drug addiction, or serious gastrointestinal, renal, hepatic or cardiovascular disease, tuberculosis, epilepsy, asthma (during past 5 years), diabetes, psychosis or glaucoma will not be eligible for this study.
* Subjects whose clinical laboratory test values are greater than 20% outside the normal range on retesting, the subject will not be significant.
* Subjects who have a history of allergic responses to the class of drug being tested should be excluded from the study.
* All subjects will have urine samples assayed for the presence of drugs of abuse as part of the clinical laboratory screening procedures and at each study period check-in. subjects found to have urin concentrations of any of the tested drugs will not be allowed to participate.
* Subjects should not have donated blood and/or plasma for at least thirty (30) days prior to the first dosing of the study.
* Subjects who have taken any investigational drug within thirty (30) days prior to the first dosing of the study will not be allowed to participate.
* Subjects who do not tolerate venipuncture will not be allowed to participate.
* Subjects who use tobacco in any form will not be eligible to participate in the study. Three months abstinence is require.
* Females will not be eligible to participate in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2002-06; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: So Ran Hong, M.D., Principal Investigator — Novum Pharmaceutical Research Services
Locations (1):
- Novum Pharmaceutical Research Services, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Finasteride (Test) First: Finasteride 5 mg Tablet (test) dosed in first period followed by Proscar® 5 mg Tablet (reference) dosed in second period
- Proscar® (Reference) First: Proscar® 5 mg Tablet (reference) dosed in first period followed by Finasteride 5 mg Tablet (test) dosed in second period
Period: First Intervention
Arm/Group | Finasteride (Test) First | Proscar® (Reference) First
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0
Period: Washout
Arm/Group | Finasteride (Test) First | Proscar® (Reference) First
Started | 16 | 16
Completed | 14 | 16
Not Completed | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention
Arm/Group | Finasteride (Test) First | Proscar® (Reference) First
Started | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Finasteride (Test) First | Proscar® (Reference) First | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 16 | 16 | 32
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 4 | 1 | 5
  Black | 9 | 11 | 20
  Hispanic | 2 | 4 | 6
  Asian | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 36 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Finasteride: Finasteride 5 mg Tablet (test) dosed in either period
- Proscar®: Proscar® 5 mg Tablet (reference) dosed in either period
Arm/Group | Finasteride | Proscar®
Number analyzed (Participants) | 30 | 30
ng/mL | 35.550 (10.170) | 35.393 (8.147)
Statistical Analysis 1: Comparison: Finasteride vs Proscar®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Geometric Test/Ref Ratio x 100 = 98.5, 90% CI [92.6 to 105] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUCinf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)
Description: Bioequivalence based on AUCinf
Time Frame: Blood samples collected over 36 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Finasteride | Proscar®
Number analyzed (Participants) | 30 | 30
ng*h/mL | 252.848 (97.525) | 256.783 (94.167)
Statistical Analysis 1: Comparison: Finasteride vs Proscar®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Geometric Test/Ref Ratio x 100 = 98.2, 90% CI [94.7 to 102] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 36 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Finasteride | Proscar®
Number analyzed (Participants) | 30 | 30
ng*h/mL | 247.327 (90.563) | 250.822 (87.883)
Statistical Analysis 1: Comparison: Finasteride vs Proscar®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Geometric Test/Ref Ratio x 100 = 98.4, 90% CI [94.9 to 102] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.